CLINICAL TRIAL: NCT05399888
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Efficacy, Safety, and Tolerability of BIIB080 in Subjects With Mild Cognitive Impairment Due to Alzheimer's Disease or Mild Alzheimer's Disease Dementia
Brief Title: A Study to Learn About the Safety of BIIB080 Injections and Whether They Can Improve Symptoms of Participants With Mild Cognitive Impairment Due to Alzheimer's Disease (AD) or Mild AD Dementia Between 50 to 80 Years of Age
Acronym: CELIA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 247AD201; 2022-501644-15 (Other: EU CT Number)
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment Due to Alzheimer's Disease; Alzheimer's Disease Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo Q12W (Placebo Comparator): Participants will receive BIIB080-matching placebo, intrathecal (IT) injection, once on Day 1 and then once every 12 weeks (Q12W) for up to 72 weeks, during the placebo-controlled period. Eligible participants will enter the LTE period, during which they will be randomized to receive BIIB080 high dose, IT injection, either Q12W or once every 24 weeks (Q24W) for an additional 96 weeks.
  Interventions: Drug: BIIB080; Drug: BIIB080-matching placebo
- BIIB080 Low Dose Q24W (Experimental): Participants will receive a low dose of BIIB080, IT injection, Q24W from Week 1 up to 72 weeks and BIIB080-matching placebo, IT injection, once at Weeks 12, 36, and 60 during the placebo-controlled period. Eligible participants will enter the LTE period, during which they will continue to receive BIIB080 low dose, IT injection, Q24W for an additional 96 weeks.
  Interventions: Drug: BIIB080; Drug: BIIB080-matching placebo
- BIIB080 High Dose Q24W (Experimental): Participants will receive a high dose of BIIB080, IT injection, Q24W from Week 1 up to 72 weeks and BIIB080-matching placebo, IT injection, once at Weeks 12, 36, and 60 during the placebo-controlled period. Eligible participants will enter the LTE period, during which they will continue to receive BIIB080 high dose, IT injection, Q24W for an additional 96 weeks.
  Interventions: Drug: BIIB080; Drug: BIIB080-matching placebo
- BIIB080 High Dose Q12W (Experimental): Participants will receive a high dose of BIIB080, IT injection, once on Day 1 and then Q12W for up to 72 weeks during the placebo-controlled period. Eligible participants will enter the LTE period, during which they will continue to receive BIIB080 high dose, IT injection, Q12W for an additional 96 weeks.
  Interventions: Drug: BIIB080

INTERVENTIONS:
Drug: BIIB080 — Administered as specified in the treatment arm.
  Other Names: ISIS 814907
Drug: BIIB080-matching placebo — Administered as specified in the treatment arm.
  Arms: BIIB080 High Dose Q24W; BIIB080 Low Dose Q24W; Placebo Q12W

SUMMARY:
In this study, researchers will learn more about a study drug called BIIB080. The study will focus on participants with mild cognitive impairment or mild dementia due to AD.

The main question researchers are trying to answer is if BIIB080 can slow the worsening of AD more than placebo. It will focus on what dose of BIIB080 slows worsening of AD the most.

To help answer this question, researchers will use the Clinical Dementia Rating-Sum of Boxes, also known as the CDR-SB.

* Clinicians use the CDR-SB to measure several categories of dementia symptoms.
* The results for each category are added together for a total score. Lower scores are better.

Researchers will also learn more about the safety of BIIB080.

The study will be split into 2 parts. The 1st part is the Placebo-Controlled Period. The 2nd part is the Long-Term Extension (LTE) Period. The 2nd part of the study will help researchers learn about the long-term safety of BIIB080, and how it affects the participant's daily life, thinking, and memory abilities in the longer term.

A description of how the study will be done is given below.

* After screening, participants will first receive either a low dose or high dose of BIIB080, or a placebo, as an injection into the fluid around the spinal cord (cerebrospinal fluid). A placebo looks like the study drug but contains no real medicine.
* Participants will receive BIIB080 or placebo once every 12 weeks or 24 weeks.
* After 76 weeks of treatment in the Placebo-Controlled Period, eligible participants will move onto the Extension Treatment period, which will last 96 weeks.
* In the extension period, participants who received placebo will be switched to high dose BIIB080 every 12 or 24 weeks.
* Participants may be in the study for up to 201 weeks, or about 4 years. This includes the screening and follow-up periods.
* Participants can continue to take certain medications for AD. Participants must be on the same dose of medication for at least 8 weeks before the screening period.
* After the screening period, most participants will visit the clinic every 6 weeks.

DETAILED DESCRIPTION:
BIIB080 is an investigational antisense therapy designed to target microtubule-associated protein tau (MAPT) messenger ribonucleic acid (mRNA) and prevent production of tau protein.

ELIGIBILITY:
Key Inclusion Criteria for Placebo-controlled Period:

* Must meet all the clinical staging criteria for MCI due to AD (Stage 3) or mild AD dementia (Stage 4) according to the National Institute on Aging at National Institutes of Health and the Alzheimer's Association (NIA-AA) and must have the following at Screening Visit 1:

  1. Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Delayed Memory Index score of ≤85, indicative of objective evidence of memory impairment.
  2. CDR global score of 0.5 for MCI due to AD or 0.5 or 1 for mild AD dementia
  3. MMSE score of 21 to 30 (inclusive).
  4. CDR Memory Box score of ≥0.5.
* Evidence of amyloid pathology as measured by positive emission tomography (PET) or cerebrospinal fluid (CSF) sampling.
* Must have 1 care partner who, in the Investigator's judgment, has frequent and sufficient contact with the participant (at least 10 hours/week) to be able to provide accurate information about the participant's cognitive and functional abilities.

Key Inclusion Criteria for LTE Period

* Ability of the participant and/or his/her legally authorized representative (e.g., parent, spouse, or legal guardian), where local regulations and institutional practices permit, as appropriate and applicable, to understand the purpose and risks of the study, to provide informed consent, and to authorize the use of confidential health information in accordance with national and local privacy regulations. Incapacitated individuals will not be enrolled in the EU (European Union) and other countries where local laws, regulations, and practices do not permit their inclusion.
* Participants must have completed the placebo-controlled period of the study, including the Week 76 visit.
* Participants must have taken at least 5 doses of BIIB080 or placebo during the placebo-controlled period.
* Medically able to undergo the study procedures (including LP [lumbar puncture]) and to adhere to the visit schedule at the time of study entry into the LTE period, as determined by the Investigator.
* Apart from a clinical diagnosis of AD, the participant must be in good health as determined by the Investigator, based on medical history.
* Must have 1 care partner who, in the Investigator's judgment, has frequent and sufficient contact with the participant (at least 10 hours/week) to be able to provide accurate information about the participant's cognitive and functional abilities.

Key Exclusion Criteria for Placebo-controlled Period:

* Known allergy to BIIB080 or a history of hypersensitivity to any of the inactive ingredients in the drug product.
* Previous participation in this study or previous studies with BIIB080.
* Use of non-disease-modifying AD medications (including but not limited to donepezil, rivastigmine, galantamine, tacrine, and memantine) at doses that have not been stable for at least 8 weeks prior to Screening Visit 1 and during the screening period up to Day 1.
* Use of any commercially available disease-modifying AD medications such as anti-amyloid monoclonal antibodies.
* Prior participation in any active or passive immunotherapy study targeting Aβ, unless documentation of receipt of placebo is available.
* Prior participation in any passive immunotherapy study targeting tau, unless the last administration occurred 6 months or 5 half-lives, whichever is sooner, prior to Screening or documentation of receipt of placebo is available.
* Prior participation in any study involving an investigational treatment targeting tau that is not a passive immunotherapy, unless documentation of receipt of placebo is available.
* Prior participation in a study of any other agent(s) not included in exclusion criteria 5, 6, and 7 with a purported disease-modifying effect in AD within 12 months, unless documentation of receipt of placebo is available.
* Prior participation in a study of any gene therapy with a purported disease-modifying effect in AD, unless documentation of receipt of placebo is available.
* Current use or previous use of medications with a purported disease-modifying effect in AD, outside of investigational studies.
* Any vaccination given within 10 days prior to Day -1. Coronavirus disease 2019 (COVID-19) vaccinations using RNA or deoxyribonucleic acid (DNA) technology are allowed during the study, as well as other types of immunization/vaccination/booster, except during the 10 days before and after clinic visits.
* Contraindications to having a brain magnetic resonance imaging (MRI) [e.g., MRI-incompatible pacemaker; MRI-incompatible aneurysm clips, artificial heart valves, or other metal foreign body; claustrophobia that cannot be medically managed]. If the MRI compatibility of implanted devices is unknown, the participant must be excluded from the study.
* Current enrollment or a plan to enroll in any interventional clinical study in which an investigational treatment or approved therapy for investigational use is administered within 52 weeks prior to the Baseline Visit.

Key Exclusion Criteria for LTE Period

* Any medical or psychiatric contraindication or clinically significant abnormality that, in the opinion of the Investigator, will substantially increase the risk associated with the participant's enrollment in and completion of the study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2029-01-08 (Estimated)

PRIMARY OUTCOMES:
Dose response in Change From Baseline to Week 76 on the CDR-SB | Baseline to Week 76
  The Clinical Dementia Rating (CDR) scale is a clinician-rated dementia staging system that tracks the progression of cognitive impairment in 6 categories (memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care). Each category is scored on a 5-point scale in which None=0, Questionable=0.5, Mild=1, Moderate=2, and Severe=3. The global CDR score is established by clinical scoring rules and has values of 0 (no dementia), 0.5, (questionable dementia), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia). The CDR-SB is obtained by adding the ratings in each of the 6 categories and ranges from 0 to 18 with higher scores indicative of greater impairment.

SECONDARY OUTCOMES:
Change From Baseline to Week 76 on the CDR-SB | Baseline to Week 76
  The CDR scale is a clinician-rated dementia staging system that tracks the progression of cognitive impairment in 6 categories (memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care). Each category is scored on a 5-point scale in which None=0, Questionable=0.5, Mild=1, Moderate=2, and Severe=3. The global CDR score is established by clinical scoring rules and has values of 0 (no dementia), 0.5, (questionable dementia), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia). The CDR-SB is obtained by adding the ratings in each of the 6 categories and ranges from 0 to 18 with higher scores indicative of greater impairment. Positive change from baseline indicates clinical decline.
Change From Baseline to Week 76 on the Alzheimer's Disease Cooperative Study Activities of Daily Living for Mild Cognitive Impairment (ADCS-ADL-MCI) | Baseline to Week 76
  The ADCS-ADL-MCI consists of 17 instrumental items (e.g., shopping, preparing meals, using household appliances) and 1 basic item (getting dressed). Ratings reflect caregiver observations about the participant's actual functioning and provide an assessment of change in the functional state of the participant over time. The total score ranges from 0 to 53, with lower values over time reflecting functional deterioration. Positive change from baseline indicates clinical improvement.
Change From Baseline to Week 76 on the Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog 13) | Baseline to Week 76
  ADAS-Cog13 comprises both cognitive tasks and clinical ratings of cognitive performance. The scale items capture word recall, ability to follow commands, the ability to correctly copy or draw an image, naming, the ability to interact with everyday objects, orientation, word recognition, memory, comprehension of spoken language, word-finding, and language ability, with a measure for delayed word recall and concentration/distractibility. The total score ranges from 0 to 85. An increase in score over time indicates increasing cognitive impairment. Positive change from baseline indicates clinical decline.
Change From Baseline to Week 76 on the Mini Mental State Examination (MMSE) | Baseline to Week 76
  The MMSE is a widely used performance-based test of global cognitive status. It consists of 11 tasks that assess orientation, word recall, attention and calculation, language abilities, and visuospatial functions. The scores from the 11 tests are combined to obtain the total score, which ranges from 0 to 30, with lower scores over time indicating increasing cognitive impairment. Positive change from baseline indicates clinical improvement.
Change From Baseline to Week 76 on the Modified Integrated Alzheimer's Disease Rating Scale (iADRS) | Baseline to Week 76
  iADRS is a composite and is calculated as a linear combination of total scores of ADAS-Cog13 and Alzheimer's Disease Cooperative Study Instrumental Activities of Daily Living Inventory (ADCS-iADL) that measures cognition and daily function. ADCS-iADL is calculated from a subset of questions from ADCS-ADL. Range for ADCS-iADL is 0-59 and higher scores reflect better performance. ADAS-Cog13 comprises cognitive tasks and clinical ratings of cognitive performance. Scale items capture word recall, ability to follow commands, ability to correctly copy/draw, naming, ability to interact with everyday objects, orientation, word recognition, memory, spoken language comprehension, word-finding, and language ability, with a measure for delayed word recall and concentration/distractibility. Score ranges from 0 to 85 with higher scores reflecting cognitive impairment. iADRS score range is 0-144 and higher scores indicate greater impairment. Positive change from baseline indicates clinical decline.
Change From Baseline to Week 76 on the Alzheimer's Disease Composite Score (ADCOMS) | Baseline to Week 76
  ADCOMS is a composite score comprised of ADAS-cog (4 items), MMSE (2 items) and CDR-SB (6 items). The total scores on the scale range from 0 to 1.97 with higher scores indicating greater impairment. Positive change from baseline indicates clinical decline.
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From first dose of study drug up to end of study of placebo-controlled period (up to Week 96)
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal (investigational) product, whether or not related to medicinal (investigational) product. TEAE is any AE that started or worsened on or after the administration of the first dose of study drug through the end of follow-up period. SAE is any untoward medical occurrence that at any dose results in death, in the view of investigator, places the participant at immediate risk of death (life-threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in congenital anomaly/birth defect or is medically important event.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (138):
- United States (36):
  - Xenoscience Inc., Phoenix, Arizona
  - HonorHealth Neurology, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Mary S. Easton Center for Alzheimer's Disease Research, UCLA, Los Angeles, California
  - PNS Clinical Research, LLC dba, Orange, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - Sutter Institute for Medical Research, Sacramento, California
  - University of California San Diego Medical Center, San Diego, California
  - University of California San Francisco (PARENT), San Francisco, California
  - Rocky Mountain Movement Disorders Center, PC, Englewood, Colorado
  - Charter Research, LLC, Lady Lake, Florida
  - K2 Medical Research, LLC, Orlando, Florida
  - Advent Health, Orlando, Florida
  - Conquest Research, Winter Park, Florida
  - Charter Research, LLC, Winter Park, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Brigham and Women's Hospital Department of Neurology, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Neurological Associates of Albany, PC, Albany, New York
  - Dent Neurologic Institute, Amherst, New York
  - New York University Medical Center PRIME, New York, New York
  - South Shore Neurologic Associates, P.C., Patchogue, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University, Durham, North Carolina
  - AMC Research, LLC, Matthews, North Carolina
  - NeuroScience Research Center, LLC., Canton, Ohio
  - University of Cincinnati Physicians Group, LLC, Cincinnati, Ohio
  - Butler Hospital, Providence, Rhode Island
  - Neurology Clinic, PC, Cordova, Tennessee
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - EvergreenHealth, Kirkland, Washington
  - Kingfisher Cooperative, LLC, Spokane, Washington
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Southern Neurology, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Mater Hospital Brisbane, South Brisbane, Queensland
- Belgium (4):
  - UZ Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
- Canada (8):
  - The Medical Arts Health Research Group, Kamloops, British Columbia
  - UBC Hospital, Vancouver, British Columbia
  - Medical Arts Health Research Group, West Vancouver, British Columbia
  - Recherches Neuro-Hippocampe Inc., d/b/a Ottawa Memory Clinic, Ottawa, Ontario
  - Toronto Memory Program (Neurology Research Inc.), Toronto, Ontario
  - Clinique de la Memoire de l'Outaouais, Gatineau, Quebec
  - Montreal Neurological Institute Clinical Research Unit, Montreal, Quebec
  - Jewish General Hospital - NETWORK, Montreal, Quebec
- Czechia (6):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava
  - Fakultni nemocnice v Motole, Prague
  - FORBELI s.r.o., Prague
  - Vestra Clinics s.r.o., Rychnov nad Kněžnou
- Denmark (2):
  - Ålborg Universitets Hospital, Aalborg
  - Rigshospitalet, Copenhagen
- Finland (2):
  - Itä-Suomen yliopisto, Kuopion kampus, Kuopio
  - CRST, Clinical Research Services Turku, Turku
- France (9):
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg, Bas Rhin
  - Hopital Purpan, Toulouse, Haute Garonne
  - Hôpital La Grave, Toulouse, Haute Garonne
  - Hopital Gui de Chauliac, Montpellier, Herault
  - CHU Nantes - Hopital Nord Laënnec, Saint-Herblain, Loire Atlantique
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - Hôpital Lariboisière, Paris, Paris
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen, Seine Maritime
  - Groupe Hospitalier Pitie-Salpetriere, Paris
- Germany (13):
  - Universitaetsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum Bayreuth GmbH- Hohe Warte, Bayreuth, Bavaria
  - Klinikum der Universität München, München, Bavaria
  - Neuro Centrum Science GmbH, Erbach im Odenwald, Hesse
  - Universitaetsmedizin Goettingen, Göttingen, Lower Saxony
  - Deutsches Zentrum fuer Neurodegenerative Erkrankungen (DZNE), Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Klinikum Altenburger Land GmbH, Altenburg, Thuringia
  - Charité - Campus Charité Mitte, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Katholisches Klinikum Bochum gGmbH, Bochum
- Italy (8):
  - Azienda Ospedaliera Card. G. Panico, Tricase, Lecce
  - Fondazione Istituto G.Giglio di Cefalù, Cefalù, Palermo
  - Ospedale di Arzignano, Arzignano VI, Vicenza
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliera e Universitaria di Perugia, Perugia
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Roma
- Japan (7):
  - Ehime University Hospital, Toon-shi, Ehime
  - Himeji Central Hospital Clinic, Himeji-shi, Hyōgo
  - Nippon Medical School Musashi Kosugi Hospital, Kawasaki-shi, Kanagawa
  - Yokohama City Minato Red Cross Hospital, Yokohama, Kanagawa
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Tokyo Metropolitan Institute for Geriatrics and Gerontology, Itabashi-ku, Tokyo-To
- Brain Research Center Amsterdam, Amsterdam, Netherlands
- Poland (10):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - PROMENTE Sp. z o.o., Bydgoszcz
  - Nzoz Novo-Med, Katowice
  - Care Clinic Centrum Medyczne, Katowice
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - SPZOZ Centralny Szpital Kliniczny UM w Lodzi, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie Kliniczny Oddział Neurologii Oddział Udarowy, Lublin
  - Centrum Medyczne Senior, Sopot
  - NeuroProtect Sp. z o.o., Warsaw
  - Mazowiecki Szpital Wojewódzki w Warszawie Sp z oo, Warsaw
- Spain (10):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - CAE Oroitu, Getxo, Vizcaya
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Fundacio ACE, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitari de Santa Maria, Lleida
  - Hospital Victoria Eugenia, Seville
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Mölndal Sjukhus, Mölndal
  - Karolinska universitetssjukhuset - Huddinge, Stockholm
- Switzerland (4):
  - Ospedale Regionale di Lugano, Lugano, Canton Ticino
  - Spitalzentrum Biel, Biel/Bienne
  - Hôpitaux Universitaires de Genève - HUG- Centre de la mémoire, Bâtiment A1 - Morier, Geneva
  - Kantonsspital St. Gallen, Sankt Gallen
- United Kingdom (11):
  - Institute of Psychiatry, Psychology and Neuroscience, London, Greater London
  - Re:Cognition Health Ltd (London), London, Greater London
  - Charing Cross Hospital, London, Greater London
  - The National Hospital for Neurology and Neurosurgery Centre, London, Greater London
  - Greater Manchester Mental Health NHS Foundation Trust, Manchester, Greater Manchester
  - Southampton General Hospital, Southampton, Hampshire
  - Warneford Hospital, Oxford, Oxfordshire
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - NeuroClin Limited, Motherwell, Strathclyde
  - Re:Cognition Health - Birmingham, Birmingham, West Midlands
  - Re Cognition Health Bristol, Bristol

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/